CLINICAL TRIAL: NCT05768334
Title: Efficacy and Tolerability of Lubiprostone in Patients With Nonalcoholic Fatty Liver Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Helwan University (Other)
Responsible Party: Principal Investigator, Mohamed El Kassas, Professor and chief of Endemic Medicine Department, Helwan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-2020
Record Dates: First submitted 2023-03-02; First posted 2023-03-14 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Lubiprostone

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lubiprostone (Active Comparator): 50 patients
  Interventions: Drug: Lubiprostone 24Mcg Oral twice daily
- Control arm (Placebo Comparator): 50 patients
  Interventions: Drug: Lubiprostone 24Mcg Oral twice daily

INTERVENTIONS:
Drug: Lubiprostone 24Mcg Oral twice daily — The patients will be randomized (closed envelopes) into one of two groups:
  1. Fifty patients will receive lubiprostone 24 mcg (microgram) twice daily.
  2. Fifty patients will receive placebo twice daily (control group). All patients will be followed for 48 weeks.

SUMMARY:
Objectives To evaluate the efficacy, safety, and tolerability of lubiprostone in patients with nonalcoholic fatty liver disease (NAFLD).

This study will include 100 patients with nonalcoholic fatty liver disease (NAFLD) recruited from the specialized NAFLD outpatient's clinic in National Hepatology and Tropical Medicine Research Institute (NHTMRI).

Study design: Randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

- 1. Age from 18-65 years. 2. Cases with NAFLD suspected by abdominal ultrasound or CT. 3. Negative viral hepatitis markers (Hepatitis B surface Antigen &Hepatitis C virus Antibody).

4. Negative autoantibodies (Antinuclear Antibody). 6. Non-cirrhotic patients as diagnosed by fibroScan (F4<14.6KPa). 7. Hepatic steatosis > 5% with MRI-PDFF.

Exclusion Criteria:

* 1. History of other forms of liver disease (including viral hepatitis, autoimmune hepatitis, hemochromatosis, Wilson's disease, and alpha-1-antitrypsin disease).

  2. Alcohol intake exceeding 30 g/day in the last 10 years or exceeding 10 g/day in the previous year (Saunders et al., 1993).

  3. Child-Pugh score > 7. 4. Cirrhotic patients diagnosed by fibroScan (F4>14.6KPa) 5. Calculated Estimated Glomerular Filtration Rate (eGFR) <60 mL/min/1.73m2. 6. Pregnancy. 7. Evidence of hepatocellular carcinoma as stated by Barcelona Clinic Liver Cancer (BCLC) (Llovet et al., 2003).

  8. Contraindications to MRI: prostetic heart valves and annuloplasty rings, metallic implants, patients who have peacemaker, and contrast allergy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
MRI-PDFF (the magnetic resonance imaging-estimated proton density fat fraction). | 48 weeks
  change in fat quantification

SECONDARY OUTCOMES:
FibroScan with CAP (Controlled Attenuation Parameter) | 48 weeks
  change in fat quantification

CONTACTS AND LOCATIONS:
Locations (1):
- National Hepatology and Tropical Medicine Research Institute, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] El-Kassas M, Mostafa H, Abdellatif W, Shoman S, Esmat G, Brahmania M, Liu H, Lee SS. Lubiprostone Reduces Fat Content on MRI-PDFF in Patients With MASLD: A 48-Week Randomised Controlled Trial. Aliment Pharmacol Ther. 2025 Feb;61(4):628-635. doi: 10.1111/apt.18478. Epub 2025 Jan 2. PMID 39744921